CLINICAL TRIAL: NCT06436326
Title: The Impact of Continuous Glucose Monitoring on Maternal and Infant's Outcomes in Gestational Diabetes: Testing the Moderating Effects of Socioeconomic and Cultural Factors
Brief Title: The Impact of Continuous Glucose Monitoring on Maternal and Infant's Outcomes in Gestational Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202311035RINC
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes Mellitus; Continuous Glucose Monitoring
Keywords: Gestational Diabetes Mellitus; Continuous Glucose Monitoring; Health Interventions
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Controlled group-Blood glucose meters (BGM) group (Other): The participants will receive structured questionnaires and blood tests (glycated albumin, fasting plasma glucose, insulin, total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein) at 24-32 weeks of pregnancy, 35 weeks of pregnancy to before delivery, and 4-12 weeks postpartum, respectively.
  Participants are required to use blood glucose meters (BGM) at "24-32 weeks of pregnancy" and "33 weeks to before delivery". After 14 days of glucose monitoring at "24-32 weeks of pregnancy", a glucose monitor report will be given to the participants. After the 14 days of glucose monitoring at "33 weeks to before delivery ", another glucose monitor report will be given to the participants.
  Interventions: Other: Blood glucose meters (BGM)
- Experimental group1-Continuous glucose monitoring (CGM) group (Experimental): The participants will receive structured questionnaires and blood tests (glycated albumin, fasting plasma glucose, insulin, total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein) at 24-32 weeks of pregnancy, 35 weeks of pregnancy to before delivery, and 4-12 weeks postpartum, respectively.
  Participants will receive a set of continuous glucose monitor (CGM) respectively at "24-32 weeks of pregnancy (first set)" and "33 weeks of pregnancy to before delivery (second set)".
  Interventions: Device: Continuous glucose monitor
- Experimental group2-Continuous glucose monitoring (CGM) with nursing care group (Experimental): The participants will receive structured questionnaires and blood tests (glycated albumin, fasting plasma glucose, insulin, total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein) at 24-32 weeks of pregnancy, 35 weeks of pregnancy to before delivery, and 4-12 weeks postpartum, respectively.
  Participants will receive a set of continuous glucose monitor (CGM) respectively at "24-32 weeks of pregnancy (first set)" and "33 weeks of pregnancy to before delivery (second set)".
  Participants will receive perinatal nursing care for gestational diabetes.
  Interventions: Device: Continuous glucose monitor; Behavioral: Perinatal nursing care for gestational diabetes

INTERVENTIONS:
Device: Continuous glucose monitor — Participants will receive a set of continuous glucose monitor (CGM) at "24-32 weeks of pregnancy (first set)" and "33 weeks of pregnancy to before delivery (second set)," respectively.
  CGM wearing instruction will be provided before the first wearing at "24-32 weeks of pregnancy". After completing the first wearing (approximately 14 days after starting to wear), the investigators will provide a glucose monitor report. The second CGM was worn from the 33rd week of pregnancy to before delivery, and another glucose monitor report was given approximately 14 days after starting to wear.
  Other Names: Abbott FreeStyle Libre 2 (CGM)
  Arms: Experimental group1-Continuous glucose monitoring (CGM) group; Experimental group2-Continuous glucose monitoring (CGM) with nursing care group
Behavioral: Perinatal nursing care for gestational diabetes — Individual nursing care and consultation for pregnant women with gestational diabetes mellitus, including glucose monitor suggestions, dietary suggestions, emotional support, breastfeeding support.
  Arms: Experimental group2-Continuous glucose monitoring (CGM) with nursing care group
Other: Blood glucose meters (BGM) — Participants are required to use blood glucose meters (BGM) at "24-32 weeks of pregnancy" and "33 weeks to before delivery". After 14 days of glucose monitoring at "24-32 weeks of pregnancy", a glucose monitor report will be given to the participants. After the 14 days of glucose monitoring at "33 weeks to before delivery ", another glucose monitor report will be given to the participants.
  Arms: Controlled group-Blood glucose meters (BGM) group

SUMMARY:
This study will discuss the impact of continuous glucose monitoring on maternal and infant's outcomes in gestational diabetes mellitus, and test the moderating effect of socioeconomic and cultural factors (dietary habits, socioeconomic status and income).

DETAILED DESCRIPTION:
Background: The global prevalence of gestational diabetes mellitus is increasing. To reduce the negative impact of gestational diabetes mellitus on maternal and fetal health, managing blood glucose during pregnancy is important, which also shows the importance of blood glucose monitoring. Continuous glucose monitoring (CGM) is different from traditional blood glucose meters (BGM). Continuous glucose monitoring is now known to have good control effects in type 1 and type 2 diabetes mellitus. However, there are still few randomized controlled trials for gestational diabetes mellitus and there are not consistent results. In addition, blood glucose management conditions vary among groups with different dietary habits, socioeconomic status and income. Food culture of Taiwan is diverse and it is easy to consume sugar or high carbohydrate foods. Continuous glucose monitoring can be more sensitive to measure glucose fluctuations, but it is still unknown whether it will have different maternal and infant health effects for groups whose glucose is prone to exceed the target range.

Objective: To explore the impact of continuous glucose monitoring on the health outcomes of mothers and infants with gestational diabetes mellitus, and to test the moderating effect of socioeconomic and cultural factors (dietary habits, socioeconomic status and income) on the relationship between continuous glucose monitoring and the health outcomes among mothers with gestational diabetes mellitus and their infants.

Methods: This study was a randomized controlled trial. It was expected that 120 pregnant women with gestational diabetes mellitus would be randomly assigned to the " Control group" (40 people) using blood glucose meters (BGM), or the "experimental group" (80 people) using continuous glucose monitoring (CGM) at a ratio of 1:2. In the "experimental group", they would be assigned to the " Experimental group1-Continuous glucose monitoring (CGM) group" (40 people) or the " Experimental group2-Continuous glucose monitoring (CGM) with nursing care group" (40 people). The " Experimental group2-Continuous glucose monitoring (CGM) with nursing care group " would provide nursing intervention during the perinatal period. The outcome variables of the three groups would be tracked and compared with 3 time points, which were 24 to 32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, and 4 to 12 weeks after delivery. The primary outcomes were maternal glycemic parameters, cardiometabolic risk factors, and fetal macrosomia. Secondary outcomes included gestational weight, depression and infant growth curve.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Pregnant women diagnosed with gestational diabetes mellitus
* Those who are willing to participate in this study

Exclusion Criteria:

* Those who have been diagnosed with diabetes mellitus "before pregnancy"
* Those whose skin is likely allergic to some materials such as tapes (signs and symptoms such as redness, swelling, itching, painful, presenting blisters or rashes caused by wearing breathable tapes, patches, etc.)
* Those who is with abnormal coagulation function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The participants of this study are pregnant women with gestational diabetes mellitus.
Enrollment: 120 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal Oral glucose tolerance test | 24-32 weeks of pregnancy, 4-12 weeks postpartum
  Oral glucose tolerance test (OGTT) including fasting, 1-hour, and 2-hour glucose levels.
Maternal glycated albumin | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  glycated albumin
Maternal albumin | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  albumin
Maternal fasting plasma glucose | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  fasting plasma glucose
Maternal insulin | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  insulin
Total cholesterol | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  total cholesterol
Triglycerides | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  triglycerides
High-density lipoprotein | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  high-density lipoprotein
Low-density lipoprotein | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  low-density lipoprotein
Fetal macrosomia | 4-12 weeks postpartum
  Fetal macrosomia is defined as a birth weight ≥4,000 g.

SECONDARY OUTCOMES:
Gestational weight gain | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery
  Gestational weight gain will be based on pre-pregnancy Body Mass Index (BMI) and classified according to the Institute of Medicine (IOM) recommendations.
Depression | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  Edinburgh Postnatal Depression Scale (EPDS) The EPDS is a 10-item questionnaire. Each item scores from 0-3. The total score is found by adding together the scores for each of the 10 items. The minimum is 0 and the maximum is 30. Scoring above 12 or 13 are likely to be suffering from depression.
Infant growth curve | 4-12 weeks postpartum
  infant growth curve
Maternal average fasting plasma glucose | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  average fasting plasma glucose
Maternal average plasma glucose, Post-cibum | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  average plasma glucose, Post-cibum
Postpartum weight retention | 4-12 weeks postpartum
  the weight change from pre-pregnancy to a period postpartum
Insulin medications | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  dosage and insulin form
Hypertensive disorders in pregnancy | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery
  Number of Participants with preeclampsia-eclampsia or gestational hypertension
Cesarean Section | 4-12 weeks postpartum
  Number of Participants with Cesarean Section
Exercise Frequency | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  Number of exercises per week.
Health behavior change of glycemic control Scale | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  A 3-item Likert scale based on the Transtheoretical model, including self-monitoring of glucose level, diet and physical activity. Each item scores from 0-4. A higher score means closer to the action or maintenance stage.
Health Belief of glycemic control Scale | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  A 21-item Likert scale based on the Health Belief model includes 5 categories: perceived susceptibility, perceived severity, perceived benefits, perceived barriers and self-efficacy.
  Each item scores from 0-4. A higher score means higher the individual's beliefs about preventing diseases or maintaining health in perceived susceptibility, perceived severity, perceived benefits and self-efficacy categories. A higher score means higher the individual's barriers to preventing diseases or maintaining health in the perceived barriers category.
Quality of life assessment | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum
  World Health Organization Quality-of-Life Scale:BREF Taiwan Version The scale evaluates four domains of quality of life ("Physical Health," "Psychological Health," "Social Relationships," and "Environment"), and contains four other questions :overall perception of quality of life, general health, dietary ,feel respected. Every domain scores from 4-20. Higher scores mean a better quality of life.
Glucose monitoring satisfaction Scale | 33 weeks of pregnancy to before delivery
  Satisfaction of using continuous glucose monitoring (CGM) or blood glucose meters (BGM) access by Likert scale. A 4-item Likert scale includes 4 categories: ease of use, painful, convenience and overall satisfaction. Each item scores from 1-5. A higher score means lower satisfaction.
Perceived benefits and barriers of CGM | 33 weeks of pregnancy to before delivery
  Benefits of CGM (BenCGM) and Burdens of CGM (BurCGM) Questionnaires. A 16-item Likert scale includes 2 categories: benefits of CGM and burdens of CGM. Each item scores from 1-5. A higher score means a higher benefit in benefit of CGM category. A higher score means higher burdens in burdens of CGM category.

CONTACTS AND LOCATIONS:
Overall Officials: HUNG-HUI CHEN, PhD, Principal Investigator — National Taiwan University Hostiptal
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch BioMedical Park Hospital, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No